CLINICAL TRIAL: NCT02838381
Title: Study of Genetic and Cellular Immunological Parameters Predictive of Disease-free Survival in Patients With Metastatic Cancer
Acronym: Epitopes-CRC01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2011/117
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Additional biological samples (Other): Additional blood samples will be realized at the inclusion of patients. Two optional blood samples could be realized if necessary with at least 3 months apart.
  Peripheral Blood Mononuclear Cells (PBMC) will be collected. Tissue tumor will be collected if available.
  Interventions: Other: Additional biological samples

INTERVENTIONS:
Other: Additional biological samples — blood and tissue samples

SUMMARY:
The aim of this study is to characterize the genetic and cellular immunological parameters of metastatic digestive cancer patients having short and long responses to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

For all patients:

* signed written informed consent

For cohort A:

* patient with metastatic colorectal cancer with first-line therapy by chemotherapy +/- surgery and with a disease-free survival > or = at 20 months
* Ct-scan realized in the previous 4 weeks and showing no progression according to the Recist criteria v1.1

For cohort B:

* patient treated for metastatic colorectal cancer and chemotherapy responder (obtention of an objective response according to the Recist criteria V1.1 in first-line therapy), with a disease-free survival < 10 months (disease progression must be confirmed by CT scan evaluation according to Recist v1.1 criteria)

For cohort C:

* patients with no metastatic rectum cancer in complete remission after chemotherapy and/or radiotherapy

For cohort D:

* patients with metastatic or locally advanced cancer in complete remission after treatment, non eligible in the other cohorts

Exclusion Criteria:

For all patients:

* patient with any medical or psychiatric condition or disease which would make the patient inappropriate for entry into this study
* patient with a neurodegenerative disease
* patient under guardianship, curator or under the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2012-06; Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
frequency of peripheral T cell immune responses in the presence of antigenic peptides associated with digestive cancer | at inclusion
progression-free survival | within 5 years after the inclusion
  time interval between the date of inclusion and the date of first progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Hôpital Nord Franche Comté, Montbéliard

REFERENCES:
- [Derived] Lopez M, Spehner L, Andre F, Viot J, Seffar E, Marguier A, Curtit E, Meynard G, Dobi E, Ladoire S, Boidot R, Loyon R, Derangere V, Bidard FC, Borg C, Mansi L, Kroemer M. Exploring the role of ESR1 mutations in metastatic hormone receptor-positive breast cancer T cell immune surveillance disruption. Breast Cancer Res. 2025 Feb 7;27(1):19. doi: 10.1186/s13058-025-01962-6. PMID 39920833